CLINICAL TRIAL: NCT04989491
Title: Multicenter Randomized Two Arms Study Evaluating the Efficacy of Prophylactic Rituximab in Adult EBV Negative Kidney Transplant Recipients on Incidence of EBV Primary Infection and Post-transplant Lymphoproliferative Disorders
Brief Title: Evaluation of the Efficacy of a Treatment by One Single Dose of Rituximab (375mg/m2 ) in the Prevention of the Epstein Barr Virus (EBV) Primary Infection and Post-transplant Lymphoproliferative Disorder in Adult EBV Seronegative Patients Who Received an EBV Seropositive Kidney Allograft
Acronym: REPLY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7678
Record Dates: First submitted 2021-07-15; First posted 2021-08-04 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Epstein-Barr Virus Infections
MeSH Terms: conditions — Epstein-Barr Virus Infections | interventions — Rituximab; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Prophylactic treatment with Rituximab: one single dose of 375mg/m2 intravenous 7 days before transplantation in case of living donor or at time of transplantation (D0 or D1) in case of transplantation with a deceased donor.
  Interventions: Drug: Rituximab
- control group (Active Comparator): Immunosuppression treatment will be given according to the practice of the centers; use of Thymoglobuline is strongly discouraged because of EBV seronegativity and risk of lymphoma. Basiliximab is recommended for induction therapy. Recommended maintenance immunosuppression consists in a calcineurin inhibitor (tacrolimus or ciclosporine), MMF and Steroids
  Interventions: Other: control group

INTERVENTIONS:
Drug: Rituximab — One single dose of rituximab intravenously (IV)
  Arms: Experimental group
Other: control group — No treatment
  Arms: control group

SUMMARY:
Epstein Barr virus infects over 90% of human population and persists during lifetime. After infecting B lymphocytes, EBV remains latent in memory B cells. In immunocompromised patients, primary infection could lead to an uncontrolled EBV infected B cells proliferation because of impaired T cell specific cytotoxicity. The latent EBV infection is characterized by expression of restricted latent gene products, which drive cell proliferation and progression to PTLD. As a consequence, EBV seronegativity and EBV mismatch are major risk factors for developing PTLD. The investigators reported in a previous work from the French Registry that the incidence of PTLD was multiplied by ten in adult EBV negative kidney transplant recipients. Moreover, even if the event is relatively rare after transplantation, the prognosis is severe with high morbidity and an overall mortality rate around 50%.

Nowadays, few and inconsistent data exist regarding beneficial preventing strategies like antiviral therapy, reduction of immunosuppression or immunoglobulin infusion in this high-risk population of EBV negative recipients. Therefore, an efficient and safe preventive treatment is still lacking to decrease PTLD incidence.

Rituximab, has been already proposed in stem cell transplant recipients as a preemptive therapy in patients with a persistent EBV viremia independently of their EBV status. A pilot study was performed in EBV negative kidney transplant recipients but in a very small population. Schachtner60 reported the cases of 5 EBV negative recipients receiving kidney from EBV positive donors after a treatment with Rituximab. Only 2 patients showed a seroconversion and no patients developed neither a viremia nor a PTLD after 49 months of follow-up.

The main objective of the investigators study is to evaluate the efficacy of early infusion of Rituximab in the prevention of EBV primary infection and post-transplant lymphoproliferative disorder (PTLD) occurrence in adult EBV negative kidney transplant recipients transplanted with an EBV positive donor.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years at transplantation)
* Kidney and kidney pancreas simultaneous transplantation
* EBV seronegative patients (IgG anti EBNA, IgG anti VCA and IgM anti VCA negative) (from 6 months before transplantation to the day of transplantation, included)
* Patient who have given written informed consent
* Negative pregnancy test and use of contraception during all the study
* EBV positive donor
* Patient affiliated to a social security scheme

Exclusion criteria:

* Patient with known HBV active infection
* Allergy to Rituximab
* Severe Immune deficiency
* Severe cardiac insufficiency
* Pregnant or lactating women
* Women of child bearing potential unless they are using a birth control method
* Patient under judicial protection or under guardianship
* Patient currently participating in another clinical trial investigating drugs. Observational studies are not considered as an exclusion criterion
* Any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, is incompatible with the participation in the study
* Unlikely to comply with the visits scheduled in the protocol.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary EBV infection | 1 year post-transplantation
  Infection assessed by a positive blood EBV viral load and/or EBV seroconversion and/or occurrence of a post-transplant lymphoproliferative disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No